CLINICAL TRIAL: NCT06084702
Title: Kids Rehydration During Exercise
Brief Title: Children Rehydration During Exercise
Acronym: ROAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Kraft Heinz Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: FP00036850
Record Dates: First submitted 2023-08-23; First posted 2023-10-16 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Dehydration in Children
MeSH Terms: interventions — Fluid Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Crossover
Who Masked: Participant
Masking Description: non-identifiable bottles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water (Placebo Comparator): Plain Water
  Interventions: Other: Rehydration with plain water
- Low Carb drink (Experimental): Roaring Water
  Interventions: Other: Rehydration Drink

INTERVENTIONS:
Other: Rehydration with plain water — Plain water without calories, sweetener, or electolytes
  Arms: Water
Other: Rehydration Drink — Roaring Water. An electrolyte drink with low Carbohydrate content
  Arms: Low Carb drink

SUMMARY:
The low fluid intake in combination with a high intake of sugar-sweetened beverages (SSB) by children is a significant concern among public health professionals. Therefore reformulation of existing commercially available beverages has been suggested as one of the strategies to change SSB beverage behaviors of children. It has been suggested that lack of flavor in plain water is one of the factors of low water intake in children. Therefore, the addition of a flavor to a low-carbohydrate beverage might increase and facilitate the voluntary fluid intake in children, and result in more effective rehydration during and after exercise. The present study aims to examine if a lower sugar flavored water will improve voluntary hydration in children that perform multiple exercise bouts within a period of 3 hours.

DETAILED DESCRIPTION:
Subject will enter a warm room with a temperature between 28-30°C (80-85°F). Then, subjects will undergo a 3-hour walk, cycle, and rest protocol. The exercise intensity is based on 70% of the subject's predicted heart rate using the formula: 220 beats per minute (bpm) - 10 years of age = 210 bpm, and 70% equals 147 bpm). This is an intensity in which the subject has an elevated breathing frequency but can still talk. During the 3-h period subject will complete the following one-hour test three times:

* 10 min walking on the treadmill at 70% of predicted max heart rate (~147 bpm)
* 5 min rest
* 10 min cycling on the cycle ergometer at 70% of predicted max heart rate (~147 bpm)
* 35 min rest

During the 3-h period, subjects will have free access to fluids Body weight and urine samples will be collected during the experiement

ELIGIBILITY:
Inclusion Criteria:

* Girls and boys age 8 to 10 years
* Willing to walk and cycle in a warm environment (80-85°F)
* Body weight ≤85th percentile for their age group

Exclusion Criteria:

* History of conditions known to alter body water balance (diabetes, renal disease, etc.)
* Drugs that (may) influence hydration status (including Selective serotonin reuptake inhibitor (SSRI), ADHD medication, diuretics and corticoids)
* Physical or mental disabilities that would prevent participation in moderate-intensity treadmill walking/jogging and cycling
* Previous diagnosis of heat stroke
* Body weight ≥86th percentile for their age group

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2023-10-14 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-04-06 (Actual)

PRIMARY OUTCOMES:
Fluid intake during the 3 hour period | 1, 2, and 3 hours of the protocol
  ad-libitum fluid intake
Net Fluid Balance based on body weight changes | 1, 2, and 3 hours of the protocol

SECONDARY OUTCOMES:
Urine output | 1, 2 and 3 hour of the protocol
  Cumulative urine volume
urine osmolality | 1, 2, and 3 hour
Urine osmotic excretion | 1, 2, and 3 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Interdisciplinary Science and Technology Building 8, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No